CLINICAL TRIAL: NCT00795678
Title: Clinical Study to Assess Entry of Chemotherapeutic Agents Into Brain Metastases in Women With Breast Cancer
Brief Title: Chemotherapeutic Agents in Brain/Breast
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE4107; P30CA043703 (NIH); CASE 4107 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Capecitabine; Cyclophosphamide; Doxorubicin; Gemcitabine; Lapatinib; Paclitaxel; Vinorelbine; Trastuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood before and after chemotherapy is administered and before and after resection of tumor in the operating room. Analysis of small portions of the brain tumor obtained at the time of craniotomy for drug collection.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — Capecitabine is an oral prodrug of 5 deoxy-5-fluorouridine (5DFRU) that is converted to 5-fluorouracil (5-FU). 5-FU is metabolized to 5-fluoro-2-deoxyuridine monophosphate (fDUMP) and 5-fluorouridine triphosphage (FUTP) which cause cell injury. Capecitabine is supplied in 150 mg (light peach colored) and 500 mg tablets (film coated)and will be administered pre-operatively.
  Other Names: Capecitabine (Xeloda®) (NSC-712807)
Drug: cyclophosphamide — Cyclophosphamide is biotransformed principally in the liver to active alkylating metabolites that cross-link tumor cell DNA. Cyclophosphamide is supplied in 100 mg, 200 mg, 500 mg and 1 gram and 2 gram vials as a white powder. The drug should be reconstituted with Sterile Water for Injection, USP, and may be diluted in either normal saline or D5W. Cyclophosphamide will be mixed in 250 mL of D5W and infused over 30 minutes prior to surgery.
  Other Names: Cyclophosphamide (Cytoxan) (NCS-26271)
Drug: doxorubicin hydrochloride — Doxorubicin is an anthracycline anticancer agent which mediates tumoricidal effects by intercalating into double-stranded DNA and producing structural changes that disrupt DNA and RNA synthesis. Doxorubicin is supplied in 10, 20, and 50 mg single use vials, and 150 mg multidose vials as a red-orange, lyophilized power which has a storage stability of a least two years. The dose will be given 60mg/m2 over 15 minutes of time pre-operatively.
  Other Names: Doxorubicin (Adriamycin) (NSC-123127)
Drug: gemcitabine hydrochloride — Gemcitabine is a fluorinated deoxynucleoside prodrug which disrupts DNA synthesis and induces apoptosis in a broad number of human tumors, including breast cancer. Gemcitabine is supplied as a lyophilized powder in sterile vials containing 200 mg of 1000 mg (1 gram) of gemcitabine as the hydrochloride salt (expressed as the free base) mannitol and sodium acetate. Dosage will be 1250mg/m2, IV pre-operatively over 30 minutes.
  Other Names: Gemcitabine (Gemzar®) (NSC-613327)
Drug: lapatinib ditosylate — : Lapatinib ditosylate monohydrate tablets, 250 mg, are oval, biconvex, orange, film-coated tablets with one side of the tablet plain and other side of the tablet embossed with FG HLS. Lapatinib may also be supplied as oval, biconvex, tan tablets, with no markings. Lapatinib will be administered for at least 3 days pre-operatively at 1250mg.
  Other Names: Lapatinib (Tykerb®) GW572016
Drug: paclitaxel — Paclitaxel will be given as an intravenous infusion (80mg/m2) the morning of surgery as specified in the protocol, diluted in 0.9% Sodium Chloride Injection, USP, or 5% Dextrose Injection. Paclitaxel will be administered via an infusion control device (pump) using non-PVC tubing and connectors, such as the IV administration sets (polyethylene or polyolefin) which are used to infuse parenteral nitroglycerin.
  Other Names: Paclitaxel (Taxol®) (NSC-673089)
Drug: vinorelbine ditartrate — Vinorelbine (Navelbine®) is a unique semi-synthetic vinca alkaloid 3', 4-didehydro-4' deoxy-C'-norvincaleukoblastine (ditartrate) (IUPAC). The pyogen free, sterile parenteral dosage form is supplied in 10 mg/1 ml ampules/vials and 50 mg/5 ml vials. It will be administered at a dosage of 25mg/m2 IV over 10-30 minutes pre-operatively.
  Other Names: Vinorelbine (Navelbine®) (INSC-608210)
Drug: Trastuzumab — Trastuzumab is a monoclonal immunoglobulin G1 kappa antibody which acts as a mediator of antibody-dependent cellular cytotoxicity (ADCC) agent through its high affinity, high specificity binding to extracellular domain of HER2 Receptor. Trastuzumab is supplied as a lyophilized, sterile powder containing 440 mg trastuzumab per vial under vacuum. Each carton contains one vial of 440 mg trastuzumab and one 30 ml vial of bacteriostatic water for injection, USP, 1.1% benzyl alcohol. This will be given the morning of surgery at 2mg/m2 IV over 90 minutes.
  Other Names: Trastuzumab (Herceptin®) (NSC #688097)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Studying samples of tumor tissue and blood from patients may help doctors understand how well these drugs can be carried to the brain.

PURPOSE: More definitive knowledge of the penetration of chemotherapeutic and other agents into the brain is necessary for the future rational design of drug and drug regimens that target brain metastases. This clinical trial is studying how well capecitabine, cyclophosphamide, doxorubicin, gemcitabine, lapatinib, paclitaxel, trastuzumab, or vinorelbine penetrates brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the concentration of capecitabine, cyclophosphamide, doxorubicin hydrochloride, gemcitabine hydrochloride, lapatinib ditosylate, paclitaxel, trastuzumab (Herceptin®), or vinorelbine ditartrate in brain metastases in women with breast cancer.
* To analyze drug penetrability by modeling the relationship between drug concentration in the tumor and drug concentration in blood samples.

OUTLINE: Patients are assigned to receive 1 of the 8 agents by the patient's treating oncologist.

Patients receive a single dose of the following study drugs immediately preceding surgery: oral capecitabine; cyclophosphamide IV over 30 minutes; doxorubicin hydrochloride IV over 15 minutes; gemcitabine hydrochloride IV over 30 minutes; oral lapatinib ditosylate*; paclitaxel IV over 3 hours; trastuzumab (Herceptin®) IV over 30-90 minutes; or vinorelbine ditartrate IV over 10-30 minutes . Patients then undergo craniotomy for resection of the brain metastases.

NOTE: *Patients receive oral lapatinib ditosylate at least 3 days prior to surgery and immediately before surgery.

All patients receiving cyclophosphamide, doxorubicin hydrochloride, gemcitabine hydrochloride, paclitaxel, or vinorelbine ditartrate also receive a single dose of pegfilgrastim subcutaneously (SC) 24-48 hours after the study drug administration OR filgrastim (G-CSF) SC once daily for 10 days, beginning 24-48 hours after the study drug administration.

Blood samples are collected periodically for pharmacological studies. Tissue samples obtained at surgical resection and blood samples are used to establish cell lines and analyzed for drug concentration by HPLC, LC-MS/MS or ELISA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast carcinoma with ≥ 1 suspected or known parenchymal brain metastases for which surgical resection or biopsy is clinically indicated
* Treating oncologist must agree that the patient would derive clinical benefit from receiving ≥ 1 of the following study agents:

  * Capecitabine, cyclophosphamide, doxorubicin hydrochloride, gemcitabine hydrochloride, lapatinib ditosylate, paclitaxel, trastuzumab (Herceptin®), or vinorelbine ditartrate
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Karnofsky performance status 50-100%
* Life expectancy ≥ 3 months
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin (total) ≤ 1.5 times ULN
* AST ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for three months after completion of study treatment
* No severe NYHA class III-IV cardiac insufficiency with uncontrolled and/or unstable cardiac or coronary artery disease
* No history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits

PRIOR CONCURRENT THERAPY:

* No toxicity > grade 2 from prior chemotherapy or radiotherapy remains at the time of study entry
* At least 60 days since prior bevacizumab
* At least 4 weeks since prior cranial radiotherapy
* At least 3 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 2 weeks since prior non-cytotoxic drugs (e.g., small molecule-targeted drugs)
* No concurrent experimental therapies
* Concurrent hormone therapy and/or trastuzumab (Herceptin®) allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from a population of breast cancer patients who are to undergo clinically indicated surgical resection of one of more symptomatic brain metastasis(es) treated at the investigational centers.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Concentration of drug | Post-Op Per Sample Collection
  Serum/plasma concentrations: measured for all agents except trastuzumab by HPLC or LC-MS/MS. Trastuzumab concentrations measured by enzyme linked immunosorbent assay. Compared to tissue levels and the extent of change in serum/plasma during the surgical process will be noted.
  Tissue Concentrations: determined by HPLC/LC-MS/MS or by ELISA. The objective would be to compare tumor concentration to brain adjacent to tumor, which often has an intact BBB. The degree of BBB compromise in the specimens will be assessed through analysis of serum protein levels and hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Peereboom, MD, Principal Investigator — Case Comprehensive Cancer Center; Robert Weil, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Memorial Sloan Kettering, New York, New York
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Morikawa A, Peereboom DM, Thorsheim HR, Samala R, Balyan R, Murphy CG, Lockman PR, Simmons A, Weil RJ, Tabar V, Steeg PS, Smith QR, Seidman AD. Capecitabine and lapatinib uptake in surgically resected brain metastases from metastatic breast cancer patients: a prospective study. Neuro Oncol. 2015 Feb;17(2):289-95. doi: 10.1093/neuonc/nou141. Epub 2014 Jul 11. PMID 25015089